CLINICAL TRIAL: NCT04396626
Title: Patient Characteristics, Treatment Patterns, and Clinical Outcomes in Patients Diagnosed With HR+/HER2- Advanced/Metastatic Breast Cancer Receiving CDK4/6i + Aromatase Inhibitor (AI) Combination Therapy as Initial Endocrine-based Treatment
Brief Title: HR+/ HER2- Advanced/ Metastatic Breast Cancer Real World Treatment Patterns and Outcomes
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely discontinued due to significant data quality issues on August 26, 2021. There were no safety concerns that led to the decision to terminate.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481144; Concerto (Other: Alias Study Number)
Record Dates: First submitted 2020-04-28; First posted 2020-05-20 (Actual); Results first posted 2022-03-21 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR + /HER2- Advanced/Metastatic Breast Cancer patients in U.S.A

SUMMARY:
This is a retrospective, observational study that will document the treatment patterns and clinical outcomes of patients diagnosed with HR+/HER2- A/MBC who received CDK4/6i combination therapy with aromatase inhibitors (AI) as the initial endocrine-based therapy in the A/MBC setting.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male sex.
2. Diagnosis (confirmed by clinical review) of A/MBC, defined as breast cancer at stage IIIB, stage IIIC, stage IV or identified as having distant metastasis.
3. Age ≥18 years at A/MBC diagnosis.
4. Initiated a CDK4/6i in combination with an AI as initial endocrine-based therapy after A/MBC diagnosis on or after 2/3/2015 and before 4/1/2019.

   •Note that the date of the start of the inclusion period reflects the month that the first CDK4/6i (ie, Palbociclib) received U.S. FDA approval.
5. Evidence of ER or PR positive disease, or absence of any indication of ER and PR negative disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of ER/PR+ status as long as ER/PR- indication is not present).
6. Evidence of HER2 negative disease, or absence of any indication of HER2 positive disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of HER2- status as long as HER2+ indication is not present).

Exclusion Criteria:

1. Enrollment in an interventional clinical trial for A/MBC during the study observation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients 18 years or older, diagnosed with HR+/HER2- A/MBC who initiated CDK4/6i combination therapy with AI as the initial endocrine-based therapy on or after 2/3/2015 and before 4/1/2019.
Sampling Method: Non-Probability Sample
Enrollment: 975 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer United States, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481144

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data for this study was not collected as study was prematurely discontinued due to significant data quality issues. There were no safety concerns that led to the decision to terminate.
Groups:
- Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI): Data for participants who received CDK4/6i along with AI as initial endocrine-based therapy for advanced and metastatic breast cancer (A/MBC) as part of their routine clinical treatment, was to be accrued from the Concerto Health AI Definitive Oncology Dataset, during this retrospective observational study.
Period: Overall Study
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Started | 975
Completed | 0
Not Completed | 975
Not completed — Premature termination of study | 975

BASELINE CHARACTERISTICS:
Groups:
- Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI): Data for participants who received CDK4/6i along with AI as initial endocrine-based therapy for advanced and metastatic breast cancer as part of their routine clinical treatment, was to be accrued from the Concerto Health AI Definitive Oncology Dataset, during this retrospective observational study.
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 975
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.78 (11.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 973
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Race and ethnicity were not collected in this study. Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Different Type of Treatment Regimens
Description: Treatment regimen was defined as one or more anti-cancer agents given in combination, over a period of time.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: Data for this study was not collected as study was prematurely discontinued due to significant data quality issues. There were no safety concerns that led to the decision to terminate.
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants Who Received Different Treatment Sequence Across Lines
Description: Lines of therapy was defined as the following progression-based lines, in which a disease progression must occur for a new regimen to be interpreted as a new line of therapy. Disease progression was taken to have occurred when a pathology report or radiological scan indicated disease progression and/or there was a physician progress note consistent with that determination.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

3. Primary Outcome: Number of Participants With Start and End Dose of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

4. Primary Outcome: Duration of Treatment of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With Reason for Treatment Discontinuation of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

6. Primary Outcome: Time to Dose Discontinuation of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

7. Primary Outcome: Number of Participants With Type of Dose Adjustments of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

8. Primary Outcome: Time to First Dose Adjustment of CDK4/6 Inhibitors
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

9. Primary Outcome: Real Progression Free Survival (rwPFS)
Description: rwPFS was defined as the time from the index date to disease progression, death, or end of record or end of data availability, whichever comes first. Index date was defined as the date of A/MBC diagnosis. Disease progression was taken to have occurred when a pathology report or radiological scan indicated disease progression and/or there was a physician progress note consistent with that determination.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

10. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the index date to disease progression, death due to any cause or end of data availability, whichever comes first. Index date was defined as the date of A/MBC diagnosis. Disease progression was taken to have occurred when a pathology report or radiological scan indicated disease progression and/or there was a physician progress note consistent with that determination
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

11. Primary Outcome: Real-World Tumor Response (rwTR)
Description: rwTR was defined as the best overall response for each regimen. Responses were classified as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), not evaluable (NE), or undocumented. The date of the first positive response (CR or PR) and of the best overall response for each regimen was collected. CR: Complete resolution of all visible disease. PR: Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. SD: no change in size of visible disease. PD: Disease progression was taken to have occurred when a pathology report or radiological scan indicated disease progression and/or there was a physician progress note consistent with that determination.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

12. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: CR: Complete resolution of all visible disease. PR: Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

13. Primary Outcome: Time to First Positive Response
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

14. Primary Outcome: Duration of Response (DOR)
Description: DOR: time from first documented occurrence of response (CR or PR) until date of first documented PD or death due to underlying cancer. Participants without a PD assessment or death were censored at the data cutoff date. CR: Complete resolution of all visible disease. PR: Partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease. PD: Disease progression was taken to have occurred when a pathology report or radiological scan indicated disease progression and/or there was a physician progress note consistent with that determination.
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

15. Primary Outcome: Duration of Initial Endocrine-based Treatment
Time Frame: From the start date of the initial endocrine-based therapy to the end date of the initial endocrine-based therapy (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

16. Primary Outcome: Duration of Treatment
Time Frame: as for outcome 15
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

17. Primary Outcome: Duration of Follow-up
Time Frame: From start to end of treatment, for a maximum of 33 months (during 15 months of retrospective observation period)
Population: as for outcome 1
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: Data for this study was not collected as study was prematurely discontinued due to significant data quality issues. There were no safety concerns that led to the decision to terminate.
Arm/Group | Cyclin-dependent Kinase 4/6 Inhibitor (CDK4/6i) + Aromatase Inhibitor (AI)
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04396626/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04396626/SAP_001.pdf